CLINICAL TRIAL: NCT00320034
Title: Double-blind, Crossover, Placebo-controlled Evaluation of the Effect of Levalbuterol (R-albuterol) on Allergen Induced Airway Inflammation In Subjects With Atopic Asthma
Brief Title: Evaluation of the Effect of Levalbuterol on Allergen Induced Airway Inflammation In Subjects With Atopic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SRC 192
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
Keywords: levalbuterol; asthma; allergen provocation; airway inflammation; clinical trial
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: R-albuterol, S-albuterol

SUMMARY:
The most commonly used drug for immediate relief of symptoms of asthma is the blue puffer, albuterol or salbutamol (Ventolin). Racemic albuterol is a mixture of two forms of albuterol which are mirror images of each other i.e. R-and S- isomers. The investigational treatments are R-albuterol and S-albuterol.

R-albuterol ( levalbuterol) has been shown to have a slightly better bronchodilator effect as compared to the racemic albuterol and is well- tolerated in patients. However it is still not clear whether the S-isomer has no effect or has a harmful effect on the airways.

The purpose of this study is to compare the effects of the R- and S- isomers on allergen induced airway inflammation in subjects with mild atopic asthma. This will give us a better idea as to whether the routine use of levalbuterol is superior to racemic albuterol.

DETAILED DESCRIPTION:
The most commonly used drug for immediate relief of symptoms of asthma is the blue puffer, albuterol or salbutamol (Ventolin). Racemic albuterol is a mixture of two forms of albuterol which are mirror images of each other i.e. R-and S- isomers. The investigational treatments are R-albuterol and S-albuterol .

R-albuterol ( levalbuterol) relieves the narrowing of the bronchial air passages in the lungs and has been approved by the U.S. FDA, but is not currently licensed for use in Canada. We have obtained approval from Health Canada to use these isomers for the purpose of this study. R-albuterol has been shown to have a slightly better bronchodilator effect as compared to the racemic albuterol and is well- tolerated in patients, with only a few mild to moderate side effects (such as palpitations, diarrhoea, abdominal pain, bodyache, leg cramps and headache). However it is still not clear whether the S-isomer has no effect or has a harmful effect on the airways.

The purpose of this study is to determine the effect of this drug, levalbuterol, on the allergen-induced inflammatory response in adult subjects with asthma. Specifically, we want to look for changes in airway eosinophils by examining sputum samples and to compare the effects of the R- and S- isomers on airway inflammation. This will help us to understand whether the racemic albuterol could worsen inflammation because of the presence of the S-isomer, and this will give us a better idea as to whether the routine use of levalbuterol is superior to racemic albuterol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (medically or surgically postmenopausal or practicing an accepted form of barrier or hormonal contraception) subjects age 18-55.
* Stable, mild atopic asthma with forced expiratory volume in one second (FEV1.0) greater than 70% of predicted for age and height, and not requiring any medical treatment other than short acting inhaled beta-agonists as needed.
* No recent or significant history of cigarette smoking (no cigarettes within six months prior to entry into the study; less than 10 pack-years cumulative history of cigarette smoking).
* Peak decrease in FEV1 in both early (0-2 hour) and late (3-7 hour) allergen-provoked response of > 15% compared with the baseline (pre-allergen challenge) spirometric determination.
* Signed written informed consent to participate in the protocol; ability to return to the outpatient clinic for repeated clinic visits.
* No history of asthma exacerbations or acute intercurrent respiratory illness (viral respiratory syndrome, bronchitis, pneumonia) for a six week period preceding entry into the screening phase of the study.

Exclusion Criteria:

* Significant gastrointestinal (including hepatic), hematological, cardiovascular, cerebrovascular or other body system disorder.
* History of an acute exacerbation, or of a respiratory tract infection at any time during the past 6 weeks.
* Baseline AST or ALT (indicators of liver damage) greater than twice the upper limit of the normal range for the local laboratory.
* History of allergy or hypersensitivity to short-acting beta-agonists.
* Inability to discontinue asthma medications for the duration of the study or receipt of oral or inhaled corticosteroids or leukotriene receptor antagonist in the three weeks prior to entry into the screening phase of the study.
* Recent (within the past 2 months) or planned (within the study period) lung volume reduction surgery.
* Psychosis, alcoholism, active substance abuse, or any personality disorder which would make compliance with this protocol problematic.
* Pregnant or nursing females.
* Any other medical or social condition which, in the opinion of the investigator, could confound the interpretation of the data derived from this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The change in airway eosinophil number (% and absolute numbers) following an allergen inhalation.

SECONDARY OUTCOMES:
Changes in:
PC20 methacholine
Allergen-induced early and late asthma responses
Airway eosinophil activation (EG-2+ eosinophils)
Levels of IL-5, RANTES, and eotaxin in sputum
Expression of PLCß1 on airway eosinophils

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, Principal Investigator — Firestone Institute for Respiratory Health, St. Joseph's Healthcare

REFERENCES:
- [Background] Lotvall J, Palmqvist M, Arvidsson P, Maloney A, Ventresca GP, Ward J. The therapeutic ratio of R-albuterol is comparable with that of RS-albuterol in asthmatic patients. J Allergy Clin Immunol. 2001 Nov;108(5):726-31. doi: 10.1067/mai.2001.119152. PMID 11692096
- [Background] Handley DA, Tinkelman D, Noonan M, Rollins TE, Snider ME, Caron J. Dose-response evaluation of levalbuterol versus racemic albuterol in patients with asthma. J Asthma. 2000 Jun;37(4):319-27. doi: 10.3109/02770900009055455. PMID 10883742